CLINICAL TRIAL: NCT00112554
Title: A Phase III Randomized of Cloretazine™ (VNP40101M) and Cytosine Arabinoside (AraC) in Patients With Acute Myeloid Leukemia in First Relapse
Brief Title: Cytarabine With or Without VNP40101M in Treating Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000430677; VION-CLI-037
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2009-02

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute | interventions — Cytarabine; laromustine

ARMS (2):
- Induction therapy arm I (Experimental): Patients receive cytarabine IV continuously on days 1-3 and VNP40101M IV over 30-60 minutes on day 2 (at least 12 hours after the start of cytarabine).
  Interventions: Drug: cytarabine; Drug: laromustine
- Induction therapy arm II (Active Comparator): Patients receive cytarabine as in arm I and placebo IV over 30-60 minutes on day 2 (at least 12 hours after the start of cytarabine).
  Interventions: Drug: cytarabine; Other: placebo

INTERVENTIONS:
Drug: cytarabine — Given IV
Drug: laromustine — Given IV
  Arms: Induction therapy arm I
Other: placebo — Given IV
  Arms: Induction therapy arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine and VNP40101M, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This randomized phase III trial is studying cytarabine and VNP40101M to see how well they work compared to cytarabine alone in treating patients with relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the complete response (CR) and CR (with platelet count < 100,000/mm^3 but ≥ 20,000/mm^3 [transfusion independent for ≥ 7 consecutive days]) (CRp) rates in patients with acute myeloid leukemia in first relapse treated with cytarabine with vs without VNP40101M.

Secondary

* Compare time to progression in patients treated with these regimens.
* Compare duration of response in patients treated with these regimens.
* Compare the survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study. Patients are stratified according to age (< 60 years vs ≥ 60 years) and duration of first complete response (CR) or CR (with platelet count < 100,000/mm³ but ≥ 20,000/mm³ [transfusion independent for ≥ 7 consecutive days]) (CRp) (< 12 months vs ≥ 12 months).

* Induction therapy: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive cytarabine IV continuously on days 1-3 and VNP40101M IV over 30-60 minutes on day 2 (at least 12 hours after the start of cytarabine).
  * Arm II: Patients receive cytarabine as in arm I and placebo IV over 30-60 minutes on day 2 (at least 12 hours after the start of cytarabine).

In both arms, patients demonstrating at least 20% reduction of blasts in bone marrow (based on total cellularity and percent blasts) after course 1 may receive 1 additional course of induction therapy between days 35-60 in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp after 1 or 2 courses of induction therapy proceed to consolidation therapy.

* Consolidation therapy: Beginning 6 weeks after initial documentation of CR or CRp, patients receive 1 course of consolidation therapy, as per induction therapy, according to their randomized treatment arm. These patients may then proceed to other consolidation, maintenance, and/or intensification therapy (including stem cell transplantation) off study at the discretion of the physician.

After completion of study treatment, patients are followed monthly for 6 months, every 2 months for 6 months, and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 420 patients (280 in arm I and 140 in arm II) will be accrued for this study within 24-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia (AML)

  * Any WHO classification, excluding acute promyelocytic leukemia
  * At least 10% blasts by bone marrow aspirate and/or biopsy
* In first relapse after achieving a first complete response (CR) OR CR (with platelet count < 100,000/mm³ but ≥ 20,000/mm³ [transfusion independent for ≥ 7 consecutive days]) (CRp) that lasted ≥ 3 months but ≤ 24 months after completion of the initial induction regimen

  * Relapse confirmed by recurrence of blasts in peripheral blood, bone marrow histopathology, and/or histologically confirmed CNS or extramedullary disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Chronic hepatitis allowed

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 3 months
* No uncontrolled arrhythmias
* No uncontrolled congestive heart failure

Pulmonary

* No severe chronic obstructive pulmonary disease
* No requirement for supplemental oxygen at rest

Immunologic

* No uncontrolled active infection

  * Infections that are controlled and under active treatment with antibiotics allowed
* No evidence of invasive fungal infection by blood or tissue cultures

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No clinical evidence of another active malignancy by tumor marker, pathology, or radiologic studies
* No other severe medical condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 12 hours since prior hydroxyurea

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior treatment while in first relapse except hydroxyurea
* No other concurrent standard or investigational treatment for AML
* No concurrent disulfiram (Antabuse®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Time to tumor progression
Duration of response
Overall response
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bonny L. Johnson, RN, MSN — Vion Pharmaceuticals
Locations (62):
- United States (24):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - American Health Network - North Meridian, Indianapolis, Indiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Nevada Cancer Institute, Las Vegas, Nevada
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Medical College, Valhalla, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - U.Z. Gasthuisberg, Leuven
  - CHU Charleroi - Site Vesale, Montigny-le-Tilleul
- Canada (6):
  - Vancouver Hospital and Health Science Center, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - Capital District Health Authority Center for Clinical Research, Halifax, Nova Scotia
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- France (5):
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Edouard Herriot, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHR Hotel Dieu, Nantes
  - Hopital Haut Leveque, Pessac
- Germany (7):
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Universitaetsfrauenklinik Frankfurt, Frankfurt
  - Universitatsklinikum Heidelberg, Heidelberg
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Medizinische Klinik und Poliklinik A - Universitaetsklinikum Muenster, Münster
  - University Wurzburg, Würzburg
- Greece (2):
  - Evaggelismos Hospital, Athens
  - University of Patras Medical School, Rio Patras
- University Medical Center Groningen, Groningen, Netherlands
- Poland (5):
  - Medical University of Gdansk, Gdansk
  - Medical University of Lodz, Lodz
  - Centrum Onkologii Ziemi Lubelskiez, Lublin
  - Wojskowy Instytut Medyczny, Warsaw
  - Institute of Haematology and Blood Transfusion, Warsaw
- Serbia (3):
  - Clinical Centre of Serbia, Belgrade
  - Clinical Centre Nis, Niš
  - Clinic Centre Novi Sad, Novi Sad
- United Kingdom (6):
  - Birmingham Heartlands Hospital, Birmingham, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leicester Royal Infirmary, Leicester, England
  - King's College Hospital, London, England
  - Manchester Royal Infirmary, Manchester, England
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Result] Giles F, Vey N, DeAngelo D, Seiter K, Stock W, Stuart R, Boskovic D, Pigneux A, Tallman M, Brandwein J, Kell J, Robak T, Staib P, Thomas X, Cahill A, Albitar M, O'Brien S. Phase 3 randomized, placebo-controlled, double-blind study of high-dose continuous infusion cytarabine alone or with laromustine (VNP40101M) in patients with acute myeloid leukemia in first relapse. Blood. 2009 Nov 5;114(19):4027-33. doi: 10.1182/blood-2009-06-229351. Epub 2009 Aug 26. PMID 19710500
- [Result] Giles FJ, Stock W, Vey N, et al.: A double blind placebo-controlled randomized phase III study of high dose continuous infusion cytosine arabinoside (araC) with or without cloretazine in patients with first relapse of acute myeloid leukemia (AML). [Abstract] Blood 108 (11): A-1970, 2006.